CLINICAL TRIAL: NCT01262534
Title: Observational Epidemiological Registry to Assess the Clinical Profile in Patients With Moderate to Severe Psoriasis in Spain
Brief Title: A Study to Assess the Clinical Profile of Patients in Spain With Moderate to Severe Psoriasis.
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017545; CNTO1275PSO4013 (Other: Janssen-Cilag S.A., Spain)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Psoriasis
Keywords: Psoriasis; comorbidities, associated treatment, quality of life
MeSH Terms: conditions — Psoriasis | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- 1: Clinical profile of patients Comorbidities and associated type of treatments will be collected.
  Interventions: Other: Clinical profile of patients
- 2: Quality of Life The Quality of Life will be assessed by 2 questionnaires (SF-36 questionnaire to analyze the overall quality of life of patients and Dermatology Life Quality Index (DLQI) to analyze the quality of life of patients in dermatological terms).
  Interventions: Other: Quality of Life
- 3: Patient Preferences about treatment Patient Benefit Index (PBI) for treatment to record patient preferences regarding psoriasis treatment.
  Interventions: Other: Patient Preferences about treatment

INTERVENTIONS:
Other: Clinical profile of patients — Comorbidities and associated type of treatments will be collected.
  Groups: 1
Other: Patient Preferences about treatment — Patient Benefit Index (PBI), for treatment to record patient preferences regarding psoriasis treatment.
  Groups: 3
Other: Quality of Life — The Quality of Life will be assessed by 2 questionnaires (SF-36 questionnaire, to analyze the overall quality of life of patients, and Dermatology Life Quality Index (DLQI), to analyze the quality of life of patients, in dermatological terms).
  Groups: 2

SUMMARY:
The purpose of this study is to assess the clinical profile of patients with moderate to severe psoriasis in Spain. The primary objective is to analyze the clinical profile of patients with moderate to severe psoriasis, as defined by a set of conditions (obesity, hypertension, diabetes, abnormal amounts of lipids in the blood, cardiovascular disease, etc.) and its correlation to the patients' quality of life. The secondary objectives are to describe the demographic characteristics and habits of the patient, to evaluate the clinical characteristics of the disease, and to describe the diagnostic and therapeutic procedures being used in standard clinical practice and the patients' expectations for these therapies.

DETAILED DESCRIPTION:
This is an epidemiological, non-interventional, multi-centre, cross-sectional, retrospective, observational study to assess the clinical profile of patients with moderate to severe psoriasis in Spain. The data for each patient will be recorded only once, in one visit. During this visit the specialist will ask the patient a series of questions to describe the existence or absence of a number of conditions and their associated treatments, to record the characteristics of psoriasis experienced by the patient and the type of associated treatment. Not applicable

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Diagnosed with psoriasis at least 6 months before the visit
* Diagnosed with moderate to severe psoriasis
* Who have been treated or not for moderate to severe psoriasis
* For whom the medical history dating back at least 6 months can be accessed
* the patient's legal representative has signed informed consent, stating that the patient understands the study purpose and requirements and grants the patient consent to participate in the study

Exclusion Criteria:

* Patient diagnosed with mild psoriasis according to the dermatologist or with a skin disease other than psoriasis
* With any type of difficulty understanding the questions in the DLQI, SF-36 and PBI questionnaires
* Who and/or whose legal representative refuses to grant written, informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from hospital sites and out-patient dermatology clinics will participate under the conditions of standard clinical practice
Sampling Method: Probability Sample
Enrollment: 1042 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.